CLINICAL TRIAL: NCT02739906
Title: A Randomised, Double Blind, Three-period Cross-over Trial to Investigate Post Prandial Blood Glucose Control With Fast-acting Human Insulin HinsBet® Compared to Insulin Lispro (Humalog®) and Regular Human Insulin (Huminsulin® Normal) After Ingestion of a Standardized Meal in Subjects With Type 1 Diabetes Mellitus (T1DM)
Brief Title: A Trial to Investigate Post Prandial Blood Glucose Control With Fast-acting Human Insulin HinsBet® Compared to Insulin Lispro (Humalog®) and Regular Human Insulin (Huminsulin® Normal) After Ingestion of a Standardized Meal in Subjects With T1DM
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Adocia (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: BC3-CT021
Record Dates: First submitted 2016-04-12; First posted 2016-04-15 (Estimated); Last update posted 2016-08-18 (Estimated); Status verified 2016-08

CONDITIONS: Type 1 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Insulin Lispro; Insulin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- HinsBet® (Experimental)
  Interventions: Drug: BioChaperone Human Insulin (HinsBet®)
- Humalog® (Active Comparator)
  Interventions: Drug: Insulin Lispro (Humalog®)
- Huminsulin® Normal (Active Comparator)
  Interventions: Drug: Regular human insulin (Huminsulin® Normal)

INTERVENTIONS:
Drug: BioChaperone Human Insulin (HinsBet®) — BioChaperone Human Insulin (HinsBet®) individualised single subcutaneous injection followed by test meal intake
  Arms: HinsBet®
Drug: Insulin Lispro (Humalog®) — Insulin Lispro (Humalog®) individualised single subcutaneous injection followed by test meal intake
  Arms: Humalog®
Drug: Regular human insulin (Huminsulin® Normal) — Regular human insulin (Huminsulin® Normal) individualised single subcutaneous injection followed by test meal intake
  Arms: Huminsulin® Normal

SUMMARY:
This is a 2 centres, randomised, double blind, three-treatment, three-period cross-over trial in subjects with type 1 diabetes mellitus.

Each subject will be administered individualised single subcutaneous doses of BioChaperone Human Insulin (HinsBet®), insulin lispro (Humalog®) and regular human insulin (Huminsulin® Normal) immediately before ingesting a standardised mixed meal.

Following trial drug administration, PK and PD assessments will be carried until 6 hours after start of the standardized test meal.

The total trial duration for an individual subject will be up to 11 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subject aged 18-64 years (both inclusive).
* Type 1 diabetes mellitus (as diagnosed clinically) >= 12 months.
* Treated with multiple daily insulin injections or CSII >= 12 months.
* Current total daily insulin treatment < 1.2 (I)U/kg/day.
* Current total daily bolus insulin treatment < 0.7 (I)U/kg/day.
* BMI 18.5-28.0 kg/m^2 (both inclusive).
* HbA1c <= 9.0 % by local laboratory analysis
* Fasting C-peptide <= 0.30 nmol/L.

Exclusion Criteria:

* Known or suspected hypersensitivity to IMPs or related products.
* Type 2 diabetes mellitus.
* Previous participation in this trial. Participation is defined as randomised.
* Participation in any clinical trial within 3 months prior to this trial.
* Clinically significant abnormal haematology, coagulation, biochemistry, lipids, or urinalysis screening tests, as judged by the Investigator considering the underlying disease.
* Presence of clinically significant acute gastrointestinal symptoms (e.g. nausea, vomiting, heartburn or diarrhoea), as judged by the Investigator.
* Known slowing of gastric emptying and or gastrointestinal surgery that in the opinion of the Investigator might change gastrointestinal motility and food absorption.
* Unusual meal habits and special diet requirements or unwillingness to eat the food provided in the trial.
* Females of childbearing potential who are pregnant, breast-feeding or intend to become pregnant or are not using highly effective contraceptive methods

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2016-04; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
BG1h | 1 hour
  Blood glucose (BG) concentration 1 hour after start of intake of a standardised meal

SECONDARY OUTCOMES:
ΔBG1h | 1 hour
  Mean change from baseline of blood glucose concentration 1 hour after start of intake of a standardised meal
AUCBG,0-1h | 1 hour
  Area under the blood glucose concentration-time curve from 0-1 hour after a standardised meal
ΔAUCBG,0-1h | 1 hour
  Incremental area under the blood glucose concentration-time curve from 0-1 hour after a standardised meal
AUCIns,0-1h | 1 hour
  Area under the serum insulin concentration-time curve from 0-1 hour
Adverse Events | Up to 11 weeks
  Number of Adverse Events
Local tolerability (Number of injection site reactions) | Up to 11 weeks
  Number of injection site reactions

CONTACTS AND LOCATIONS:
Overall Officials: Oliver Klein, MD, Principal Investigator — Profil GmbH
Locations (2):
- Germany (2):
  - Profil Mainz GmbH & Co.KG, Mainz
  - Profil GmbH, Neuss